CLINICAL TRIAL: NCT01111539
Title: A Multicenter, Randomized, Double-blind Study to Evaluate the Efficacy, Safety and Tolerability of an Oral Aripiprazole/Escitalopram Combination Therapy in Patients With Major Depressive Disorder
Brief Title: Study to Evaluate the Efficacy, Safety and Tolerability of an Oral Aripiprazole/Escitalopram Combination Therapy in Participants With Major Depressive Disorder (MDD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early due to Sponsor decision, closure of this combination therapy program is unrelated to any safety issues, no signals of concern.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31-08-255; 2010-018796-21 (EudraCT Number)
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major Depressive Disorder; MDD; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase B: Single-blind Prospective Treatment Phase (Experimental): Participants received initial dose of escitalopram 10 milligram (mg) blinded capsule (over-encapsulated tablet), orally, once daily, increased to 20 mg/day at the end of Week 1 based upon tolerability profile, for up to maximum of Week 8. No dose reductions were allowed after Week 4 and no dose increments were allowed after Week 3. Participants with incomplete response at the end of the Phase B (Week 8) entered Phase C and the rest of the participants continued to Phase B+.
  Interventions: Drug: Escitalopram; Drug: Blinded capsule
- Phase B+: Single-blind Phase B Responders (Experimental): Participants with response (≥50% reduction in depressive symptom severity in Hamilton Depression Rating Scale {HAM-D17} Total Score; or a HAM-D17 Total Score of <14 at Week 8 or a Clinical Global Impression of Improvement {CGI-I} Score of <3 at the Week 6 or 8) at the end of the Phase B (Week 8) continued treatment with the single-blind escitalopram monotherapy at the dose (10 or 20 mg/day blinded capsules) taken during the final week of Phase B, for up to maximum of Week 14, in Phase B+.
  Interventions: Drug: Escitalopram; Drug: Blinded capsule
- Phase C: Aripiprazole/Escitalopram Combination (Experimental): Participants with incomplete response (less than 50% reduction in depressive symptom severity between Baseline and Week 8 measured by the HAM-D17 Total Score and HAM-D17 Total Score of ≥14 at Week 8 and CGI-I Score of ≥3 at Week 6 and 8) at Week 8 received initial dose of aripiprazole 6 mg blinded capsule, orally, once daily at Week 9. Participants were up titrated to aripiprazole target dose of 12 mg/day at Week 10 (if initial 6 mg/day dose was tolerated) or down titrated to 3 mg/day (if significant tolerability issues arise on initial 6 mg/day dose), and thereafter received same dose up to maximum of Week 14. No dose increases were allowed for aripiprazole after end of Week 12, however, doses might be decreased at any visit based upon tolerability. In combination with aripiprazole, participants received escitalopram (10 or 20 mg/day blinded capsules) taken during final week of Phase B for up to maximum Week 14, in Phase C. No dose adjustments allowed for escitalopram during Phase C.
  Interventions: Drug: Escitalopram; Drug: Aripiprazole; Drug: Blinded capsule
- Phase C: Escitalopram Monotherapy (Experimental): Participants with incomplete response (less than a 50% reduction in depressive symptom severity between the Baseline and Week 8 as measured by the HAM-D17 Total Score and a HAM-D17 Total Score of ≥14 at Week 8 and a CGI-I Score of ≥3 at Week 6 and 8) at Week 8, received escitalopram dose (10 or 20 mg/day blinded capsules) taken during the final week of Phase B for up to maximum Week 14, in Phase C. No dose adjustments were allowed for escitalopram monotherapy during Phase C.
  Interventions: Drug: Escitalopram; Drug: Blinded capsule
- Phase C: Aripiprazole Monotherapy (Experimental): Participants with incomplete response (less than a 50% reduction in depressive symptom severity between the Baseline and Week 8 as measured by the HAM-D17 Total Score and a HAM-D17 Total Score of ≥14 at Week 8 and a CGI-I Score of ≥3 at Week 6 and 8) at Week 8, received initial dose of aripiprazole 6 mg blinded capsule, orally, once daily for Week 9. Participants were up titrated to the aripiprazole target dose of 12 mg/day at Week 10 (if the initial 6 mg/day dose was tolerated) or down titrated to 3 mg/day (if significant tolerability issues arise on the initial 6 mg/day dose), and thereafter received the same dose for up to maximum of Week 14. No dose increases were allowed for aripiprazole after the end of Week 12, however, doses might be decreased at any visit based upon tolerability.
  Interventions: Drug: Aripiprazole; Drug: Blinded capsule

INTERVENTIONS:
Drug: Escitalopram — Escitalopram capsule administered orally, once daily without regard to meals.
  Arms: Phase B+: Single-blind Phase B Responders; Phase B: Single-blind Prospective Treatment Phase; Phase C: Aripiprazole/Escitalopram Combination; Phase C: Escitalopram Monotherapy
Drug: Aripiprazole — Aripiprazole capsule administered orally, once daily without regard to meals.
  Arms: Phase C: Aripiprazole Monotherapy; Phase C: Aripiprazole/Escitalopram Combination
Drug: Blinded capsule — Blinded capsule administered orally, once daily.

SUMMARY:
This will be a multicenter, randomized, double-blind study designed to assess the efficacy, safety and tolerability of an oral Aripiprazole/Escitalopram combination therapy in participants with MDD who have demonstrated an incomplete response to a prospective trial of Escitalopram, and report a treatment history for the current MDD episode of an inadequate response to at least one and no more than three adequate trials of an approved antidepressant other than Escitalopram. An inadequate response is defined as less than a 50% reduction in depressive symptom severity as assessed by the participant's self-report on the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (ATRQ) and evaluated by the investigator as part of the participant's medical and psychiatric history. An adequate trial is defined as an antidepressant treatment for at least 6 weeks duration (or at least 3 weeks for combination treatments) at an approved dose as specified in the ATRQ.

DETAILED DESCRIPTION:
The study will be organized as follows:

* Screening Phase
* Single-blind Prospective Treatment Phase
* Single-blind Continuation Phase (Responder) or Double-blind Randomization Phase (non-Responder)
* 30 day Post Treatment Follow-up

Assigned Interventions:

* Escitalopram monotherapy
* Aripiprazole/Escitalopram combination therapy
* Aripiprazole monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Participants with a current diagnosis of a major depressive episode. The current depressive episode must be ≥8 weeks in duration
* Participants willing to discontinue all prohibited psychotropic medication starting from the time of signing the informed consent and during the study period
* Participants with a Hamilton Depression Rating Scale (HAM-D17) Total Score ≥18 at the Baseline Visit for the Prospective Treatment Phase

Exclusion Criteria:

* Lack of prior treatment with an antidepressant during the current depressive episode
* Participants who report treatment with adjunctive or monotherapy antipsychotic treatment during the current depressive episode
* Participants experiencing hallucinations, delusions or any psychotic symptomatology in the current depressive episode
* Participants with epilepsy or significant history of seizure disorders
* Participants with a clinically significant current diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder
* Participants who have received electroconvulsive therapy (ECT) in the last 10 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2010-07-13 (Actual); Primary Completion 2011-09-20 (Actual); Study Completion 2011-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (56):
- United States (24):
  - Cerritos, California
  - Costa Mesa, California
  - Irvine, California
  - San Diego, California
  - Santa Ana, California
  - Denver, Colorado
  - Cromwell, Connecticut
  - Hartford, Connecticut
  - Fort Walton Beach, Florida
  - Gainesville, Florida
  - Chicago, Illinois
  - Libertyville, Illinois
  - Boston, Massachusetts
  - Fall River, Massachusetts
  - Albuquerque, New Mexico
  - Fresh Meadows, New York
  - Staten Island, New York
  - The Bronx, New York
  - Cary, North Carolina
  - Oklahoma City, Oklahoma
  - Memphis, Tennessee
  - DeSoto, Texas
  - Richmond, Virginia
  - Brown Deer, Wisconsin
- Estonia (3):
  - Jämejala
  - Tallinn
  - Tartu
- Finland (3):
  - Helsinki
  - Kuopio
  - Oulu
- Germany (4):
  - Berlin
  - Hamburg
  - Munich
  - Ostfildern
- India (6):
  - Study Site 1, Ahmedabad, Gujarat
  - Study Site 2, Ahmedabad, Gujarat
  - Mangalore, Karnataka
  - Mumbai, Maharashtra
  - Pune, Maharashtra
  - Varanasi, Uttar Pradesh
- Italy (2):
  - Catania
  - Siena
- Mexico (8):
  - Tlalnepantla, Estado Do Mexico
  - Zapopan, Jalisco
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - Culiacán, Sinaloa
  - Villahermosa, Tabasco
  - Durango
  - San Luis Potosí City
- South Korea (2):
  - Gwangju
  - Seoul
- Taiwan (4):
  - Changhua
  - Kaohsiung City
  - Keelung
  - Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 69 investigative sites in Estonia, Finland, Germany, India, Italy, Mexico, South Korea, Taiwan, Ukraine, and the United States from 13 July 2010 to 20 September 2011.
Pre-assignment Details: A total of 211 participants were enrolled in Phase B (Single-blind Prospective Treatment Phase) to receive escitalopram monotherapy(10 or 20mg/day),of which 45 responders continued to Phase B+(Single-blind Phase B Responders),received escitalopram monotherapy(10 or 20mg/day),84 non-responders were randomized in 1:1:1 ratio to Phase C(Double-blind Randomization Phase),received aripiprazole/escitalopram combination therapy or escitalopram or aripiprazole monotherapy.
Period: Phase B (Day 1 to Week 8)
Arm/Group | Phase B: Single-blind Prospective Treatment Phase | Phase B+: Single-blind Phase B Responders | Phase C: Aripiprazole/Escitalopram Combination | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy
Started | 211 | 0 | 0 | 0 | 0
Completed | 129 | 0 | 0 | 0 | 0
Not Completed | 82 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 6 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0 | 0 | 0
Not completed — Sponsor Discontinued Study | 60 | 0 | 0 | 0 | 0
Not completed — Investigator Withdrew Subject | 1 | 0 | 0 | 0 | 0
Not completed — Subject Withdrew Consent | 7 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy as Determined by the Investigator | 1 | 0 | 0 | 0 | 0
Period: Phase B+ and Phase C (Weeks 9 to 14)
Arm/Group | Phase B: Single-blind Prospective Treatment Phase | Phase B+: Single-blind Phase B Responders | Phase C: Aripiprazole/Escitalopram Combination | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy
Started | 0 | 45 | 28 | 28 | 28
Intent-to-treat (ITT) Sample (ITT Sample included all participants in the Randomized Sample who received at least one dose of double-blind study medication and had at least one post-randomization efficacy evaluation.) | 0 | 45 | 28 | 27 | 28
Safety Sample (Safety Sample included those randomized participants in Phase C who received at least one dose of double-blind study medication as indicated on the dosing record.) | 0 | 45 | 28 | 27 | 28
Completed | 0 | 38 | 22 | 20 | 18
Not Completed | 0 | 7 | 6 | 8 | 10
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 2
Not completed — Sponsor Discontinued Study | 0 | 7 | 4 | 5 | 5
Not completed — Subject Met Withdrawal Criteria | 0 | 0 | 0 | 0 | 1
Not completed — Investigator Withdrew Subject | 0 | 0 | 0 | 1 | 0
Not completed — Subject Withdrew Consent | 0 | 0 | 0 | 2 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Phase B Sample included all participants who took at least one dose of escitalopram as indicated on the dosing record.
Arm/Group | Phase B: Single-blind Prospective Treatment Phase
Number analyzed (Participants) | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140
  Male | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42
  Not Hispanic or Latino | 168
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 16
  Asian | 36
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 130
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Phase C: Mean Change From End of Phase B (Week 8) in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score to End of Phase C (Week 14)
Description: The MADRS assessed severity of depressive symptoms. It ranges from a minimum of 0 to a maximum of 60 (higher scores indicating a greater severity of depressive symptoms). Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and a lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). A negative change from Week 8 indicates improvement.
Time Frame: Week 8 to Week 14
Population: ITT Sample included all participants in the Randomized Sample who received at least one dose of double-blind study medication and had at least one post-randomization efficacy evaluation.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase C: Aripiprazole/Escitalopram Combination | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy
Number analyzed (Participants) | 28 | 27 | 28
score on a scale | -8.0 (1.5) | -7.0 (1.5) | -4.3 (1.5)
Statistical Analysis 1: Comparison: Phase C: Aripiprazole/Escitalopram Combination vs Phase C: Escitalopram Monotherapy; The statistical analyses was performed by fitting an analysis of covariance (ANCOVA) model to the change from baseline data (Week 8 Visit) for the MADRS Total Score at the Week 14 visit (LOCF). The model included baseline MADRS Total Score as a covariate and treatment as the main effect; Test type: Superiority; p = 0.644, ANCOVA; Treatment Difference = -1.0, 95% CI 2-sided [-5.2 to 3.3]
Statistical Analysis 2: Comparison: Phase C: Aripiprazole/Escitalopram Combination vs Phase C: Aripiprazole Monotherapy; The statistical analyses will be performed by fitting an ANCOVA model to the change from baseline data (Week 8 Visit) for the MADRS Total Score at the Week 14 visit (LOCF). The model will include baseline MADRS Total Score as a covariate and treatment as the main effect; Test type: Superiority; p = 0.080, ANCOVA; Treatment Difference = -3.7, 95% CI 2-sided [-7.8 to 0.4]

2. Secondary Outcome: Phase C: Mean Clinical Global Impression - Improvement (CGI-I) Scale Score at the End of Phase C (Week 14)
Description: CGI-I is a 7-point clinician-rated scale ranging from 1 to 7, rated as 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. A higher score indicates greater impairment.
Time Frame: Week 14
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Phase C: Aripiprazole/Escitalopram Combination | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy
Number analyzed (Participants) | 28 | 27 | 28
score on a scale | 2.6 (0.2) | 2.9 (0.2) | 3.0 (0.1)
Statistical Analysis 1: Comparison: Phase C: Aripiprazole/Escitalopram Combination vs Phase C: Escitalopram Monotherapy; Test type: Superiority; p = 0.366, Cochran-Mantel-Haenszel; Treatment Difference = -0.3, 95% CI 2-sided [-0.8 to 0.3]
Statistical Analysis 2: Comparison: Phase C: Aripiprazole/Escitalopram Combination vs Phase C: Aripiprazole Monotherapy; Test type: Superiority; p = 0.138, Cochran-Mantel-Haenszel; Treatment Difference = -0.4, 95% CI 2-sided [-0.9 to 0.1]

3. Secondary Outcome: Phase C: Mean Change From End of Phase B (Week 8) in the Sheehan Disability Scale (SDS) Mean Score to End of Phase C (Week 14)
Description: SDS is a 3-item clinician-rated questionnaire used to evaluate impairments in the domains of work, social life/leisure, and family life/home responsibility. The participant is asked to rate the degree to which their functioning is impaired on an 11-point scale, ranging from 0 (not at all) to 10 (extremely). The scores for the 3 domains are summed into a total score that ranges from 0 (unimpaired) to 30 (highly impaired). A higher score indicates greater impairment. A negative change from Week 8 indicates improvement.
Time Frame: Week 8 to Week 14
Population: ITT Sample included all participants in the Randomized Sample who received at least one dose of double-blind study medication and had at least one post-randomization efficacy evaluation. Overall number of participants analyzed are the participants with evaluable data for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase C: Aripiprazole/Escitalopram Combination | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy
Number analyzed (Participants) | 27 | 25 | 26
score on a scale | -1.2 (0.4) | -1.2 (0.4) | -0.2 (0.4)
Statistical Analysis 1: Comparison: Phase C: Aripiprazole/Escitalopram Combination vs Phase C: Escitalopram Monotherapy; Test type: Superiority; p = 0.995, ANCOVA; Treatment Difference = -0.0, 95% CI 2-sided [-1.2 to 1.2]
Statistical Analysis 2: Comparison: Phase C: Aripiprazole/Escitalopram Combination vs Phase C: Aripiprazole Monotherapy; Test type: Superiority; p = 0.118, ANCOVA; Treatment Difference = -0.9, 95% CI 2-sided [-2.1 to 0.2]

ADVERSE EVENTS:
Time Frame: From first dose through 30 days after last dose of study drug (up to approximately 18 weeks)
Description: Phase B Sample- participants who took at least one dose of escitalopram. Phase B+ Sample - participants who responded at end of Phase B (were therefore not randomized) and continued on single-blind escitalopram beyond Week 8. Safety Sample(SS) included those randomized participants in Phase C who received at least one dose of double-blind study medication. 1 participant randomized to escitalopram group, was withdrawn by investigator prior to dosing in Phase C and thus was not included in the SS.
Arm/Group | Phase B: Single-blind Prospective Treatment Phase | Phase B+: Single-blind Phase B Responders | Phase C: Aripiprazole/Escitalopram Combination | Phase C: Escitalopram Monotherapy | Phase C: Aripiprazole Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/211 | 0/45 | 0/28 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 2/211 | 0/45 | 0/28 | 1/27 | 1/28
Other Adverse Events (participants affected / at risk) | 82/211 | 3/45 | 18/28 | 11/27 | 17/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase B: Single-blind Prospective Treatment Phase (N=211) | Phase B+: Single-blind Phase B Responders (N=45) | Phase C: Aripiprazole/Escitalopram Combination (N=28) | Phase C: Escitalopram Monotherapy (N=27) | Phase C: Aripiprazole Monotherapy (N=28)
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase B: Single-blind Prospective Treatment Phase (N=211) | Phase B+: Single-blind Phase B Responders (N=45) | Phase C: Aripiprazole/Escitalopram Combination (N=28) | Phase C: Escitalopram Monotherapy (N=27) | Phase C: Aripiprazole Monotherapy (N=28)
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 2
Vision blurred (Eye disorders) | 2 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 12 | 1 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 8 | 1 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 21 | 0 | 1 | 2 | 4
Feeling jittery (General disorders) | 0 | 0 | 1 | 0 | 2
Irritability (General disorders) | 2 | 0 | 2 | 0 | 2
Seasonal allergy (Immune system disorders) | 2 | 0 | 0 | 0 | 3
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 1
Akathisia (Nervous system disorders) | 0 | 0 | 2 | 1 | 5
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 6 | 0 | 1 | 0 | 2
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 36 | 1 | 2 | 2 | 4
Sedation (Nervous system disorders) | 3 | 0 | 2 | 0 | 4
Somnolence (Nervous system disorders) | 12 | 0 | 3 | 3 | 1
Insomnia (Psychiatric disorders) | 4 | 0 | 3 | 2 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 4 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
The trial was terminated to allow support of additional programs in the central nervous system (CNS) therapeutic area where limited therapies are available and, thus, there exists heightened unmet medical need and is unrelated to any safety issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.